CLINICAL TRIAL: NCT00192205
Title: A Prospective, Randomized, Open-Label, Controlled Trial to Compare the Safety, Tolerability and Efficacy of Influenza Virus Vaccine, Trivalent, Type A&B, Live, Cold-Adapted (CAIV-T) With Influenza Virus Vaccine, Trivalent, Inactivated (TIV) in Children With a History of Recurrent Respiratory Tract Infections Aged 6 Months to Less Than 72 Months
Brief Title: Trial to Compare the Safety,Tolerability and Efficacy of Influenza Virus Vaccine, (CAIV-T) With Influenza Virus Vaccine, Trivalent, Inactivated (TIV) in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D153-P514
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-10

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

INTERVENTIONS:
Biological: CAIV-T or TIV

SUMMARY:
- Trial to compare the efficacy of the liquid formulation of CAIV-T with TIV against culture confirmed influenza illness in children.

DETAILED DESCRIPTION:
* The purpose of this study is to compare the efficacy of the liquid formulation of CAIV-T with TIV against culture confirmed influenza illness in children with a history of recurrent RTIs aged at least 6 months and less than 72 months of age.
* The trial also provides the opportunity to compare the efficacy of CAIV-T with TIV on acute otitis media.

ELIGIBILITY:
Inclusion Criteria:

* who are aged at least 6 months and less than 72 months of age at the time of enrolment;
* who have experienced two or more practitioner attended RTIs* in the past 12 months (since birth if less than 12 months old); * RTIs are defined as upper RTIs including (but not limited to) common cold, acute otitis media and lower RTIs including (but not limited to) bronchiolitis, bronchitis and pneumonia.
* whose parent(s)/legal guardian(s) have provided written informed consent after the nature of the study has been explained;
* who, along with their parent(s)/legal guardian(s), will be available for duration of the trial;
* whose parent(s)/legal guardian(s), can be reached by study staff for the post-vaccination contacts [telephone, clinic or home visit].

Exclusion Criteria:

* whose parent(s)/legal guardian(s) are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease;
* with Down's syndrome or other known cytogenetic disorders;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids of a dose equivalent to (i) 2mg/kg/day or greater of Prednisolone or (ii) equivalent to a total of 20 mg/day or greater for children who weigh more than 10kg, for more than 14 days duration until 2 weeks after corticosteroids have been discontinued 27;
* who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study;
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrolment through to the conclusion of the study;
* who have an immunosuppressed or an immunocompromised individual living in the same household;
* who, at any time prior to entry into this study, received a dose of any influenza vaccine (commercial or investigational) or is anticipated to receive a non-study influenza vaccine after enrollment;
* with a documented history of hypersensitivity to egg or egg protein or any other component of CAIV-T or TIV;
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to enrolment or for which use is anticipated during the study;
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results;

Note: Pregnancy in any person who has regular contact with the subject is not a contraindication to the enrolment or ongoing participation of the subject in the study.

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2200
Dates: Start 2002-10; Study Completion 2003-06

PRIMARY OUTCOMES:
To demostrate that the efficacy over one season against culture-confirmed influenza-illness caused by community-acquired subtypes antigenically similar to those contained in the vaccine

SECONDARY OUTCOMES:
To demostrate that the efficacy over one season of CAIV-T is not inferior to that of TIV against culture-confirmed influenza-illness of any subtype
To demonstrate that the efficacy of CAIV-T is not inferior to that of TIV against clinically-defined acute otitis media
To compare the rate of occurence over a defined surveillance period in children with a histroy of recurrent RTIs

CONTACTS AND LOCATIONS:
Locations (2):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- Hospital de Txagorritxu, Vitoria-Gasteiz, Spain